CLINICAL TRIAL: NCT02468219
Title: Cardiovascular RehAbilitation in Patients With Severe AoRtic StEnosis Submitted to Valvar Correction: Effects on Muscle Architecture, Tissue Oxygenation, EndoThelial Function, Inflammatory Profile, and AutoNomic Control - Randomized Trial
Brief Title: Cardiovascular Rehabilitation in Patients With Severe Aortic Stenosis Submitted to Valvar Correction
Acronym: CARE-AS-MOTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Marlus Karsten, Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR00002509/FWA
Record Dates: First submitted 2015-05-21; First posted 2015-06-10 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic stenosis; aortic valve replacement; transcatheter aortic valve implantation; frailty; cardiac rehabilitation
MeSH Terms: conditions — Aortic Valve Stenosis; Frailty

STUDY DESIGN:
Intervention Model Description: This study will be divided into four phases: phase 1 (pre-procedure rehabilitation); phase 2 (early post-procedure rehabilitation); phase 3 (late post-procedure rehabilitation), and phase 4 (follow-up).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aortic valve replacement (Active Comparator): patients with aortic stenosis submitted to aortic valve replacement procedure
  Interventions: Behavioral: cardiovascular rehabilitation program
- transcatheter aortic valve implantation (Experimental): patients with aortic stenosis who underwent to transcatheter aortic valve implantation
  Interventions: Behavioral: cardiovascular rehabilitation program

INTERVENTIONS:
Behavioral: cardiovascular rehabilitation program — Phase I: 2-weeks of respiratory muscle training and neuromuscular electrical stimulation (daily at hospital).
  Phase II: 6-weeks of respiratory muscle training and neuromuscular electrical stimulation (daily at home).
  Phase III: 8-weeks of supervised, structured, combined aerobic and resistance training.

SUMMARY:
This study will be evaluate the autonomic, endothelial and hemodynamic functions, inspiratory muscle strength, peripheral tissue oxygenation, peripheral and respiratory muscle architecture, and inflammatory profile of severe AS patients submitted undergoing to valve replacement (sAVR) or transcatheter aortic valve implantation (TAVI), and their influence on the pathophysiological mechanisms involved in cardiovascular rehabilitation.

DETAILED DESCRIPTION:
Background: Aortic stenosis (AS) is a disease characterized by the inadequate valve opening, compromising the cardiac output. Surgical aortic valve replacement (sAVR) is the procedure indicates for valve repair in AS symptomatic cases whereas the transcatheter aortic valve implantation (TAVI) is the procedure indicates for sAVR contraindicated cases.

Objective: To evaluate the effect of the cardiac rehabilitation program (pre-procedure, early post-procedure, and late post-procedure) in autonomic, endothelial and hemodynamic functions, inspiratory muscle strength, peripheral tissue oxygenation, peripheral and respiratory muscle architecture, and inflammatory profile of severe AS patients submitted to a valve repair procedure (sAVR or TAVI).

Methods: The present study will be a randomized double-blind clinical trial in patients indicated to valve repair procedure. This research will be divided into four phases: phase 1 (pre-procedure); phase 2 (early post-procedure); phase 3 (late post-procedure) and phase 4 (follow-up). Phase 1: participants will be randomized in PR-I (pre-intervention) or PR-C (control). Pre-procedure rehabilitation program will consist of daily neuromuscular electrical stimulation (NMES) in knee extensor muscles and inspiratory muscle training (IMT) sessions. PR-C group will receive daily visits, but with a NMES + IMT protocols using a minimal load. Phase 2: a new random will be done between ER-II or ER-CI (intervention) and ER-IC or ER-CC (control). Intervention groups will undertake an early post-procedure rehabilitation (NMES in knee extensor muscle plus IMT for six weeks). Control groups will receive the same protocol using a minimal load without load progression. Phase 3: all patients will be referred to the conventional cardiac rehabilitation program (aerobic and resistance training) for 8-weeks. Phase 4: follow-up (no interventions), will be done after 3, 6, 9 and 12 months. Assessment protocol will be composed by cardiopulmonary exercise test, autonomic (heart rate variability), endothelial (flow-mediated vasodilation), hemodynamic function (cardiothoracic impedance) functional capacity (six-minute walk test), maximum inspiratory pressure, peripheral and respiratory muscle architecture (ultrasonography), and tissue oxygenation (near-infrared spectroscopy), and inflammatory profile (OxLDL, TGF-β, TNF-α, IL-1b, IL-10 and ICAM-1) Appropriate statistic tests will be used to compare the time-rehabilitation (experimental vs sham) and group-interaction (sAVR vs TAVI). If samples are abandoned or lost, basal data will be double entered to characterize the intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria: patients NYHA class II-IV who has not participated in a CRP three months before recruitment; older than 40 years; of both genders; with degenerative AS and indication for valve repair. The patients will not know which protocol to undergo.

Exclusion Criteria: patients with low cognitive level to perform the assessment or intervention procedures; that exhibit unstable angina or any contraindications for the treatment or measurements; as well musculoskeletal, cerebrovascular, or psychiatric disease that prevents their participation in the research.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory function | Changes from 8 and 16 weeks
  Peak oxygen consumption (VO2PEAK), among other physiologic markers.

SECONDARY OUTCOMES:
Autonomic function | Change from 2, 8 and 16 weeks
  will be evaluated by heart rate variability using a wrist heart rate monitor following the recommendations of ESC/NASPE Task Force.
Endothelial function | Changes from 2, 8 and 16 weeks
  will be investigated by endothelium-dependent flow-mediated vasodilation (FMD) technique following the International Brachial Artery Reactivity Task Force.
Hemodynamic function | Changes from 2, 8 and 16 weeks
  will be evaluated the cardiac output using a cardiothoracic impedance device (noninvasive approach).
Inflammatory profile | Changes from 2, 8 and 16 weeks
  Plasma levels will be determined by enzyme-linked immunosorbent assay using commercial systems.
Inspiratory muscle strength | Changes from 2, 8 and 16 weeks
  Will be assessed as maximum inspiratory pressure (MIP) using a digital device following recommendations of the American Thoracic Society and European Respiratory Society.
Muscle architecture (peripheral muscles) | Changes from 8 and 16 weeks
  Will be evaluated the muscle thickness (cross-sectional area) of quadriceps using a ultrasonography system.
Muscle architecture (respiratory muscles) | Changes from 8 and 16 weeks
  Will be evaluated the diaphragm thickness (cross-sectional area) of quadriceps using a ultrasonography system.
Tissue oxygenation | Changes from 2, 8 and 16 weeks
  near-infrared spectroscopy (NIRS) will be used to verify muscle oxygenation (quadriceps and respiratory muscles).
Functional capacity | Changes from 8 and 16 weeks
  The patients under favorable clinical conditions will be functionally evaluated by the Six-Minute Walk Test (6MWT) according to current guidelines.
Mortality | Change from 3, 6 and 12 months post protocol
  to evaluate the survival rate of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Marlus Karsten, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Marlus Karsten, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Montemezzo D, Fregonezi GA, Pereira DA, Britto RR, Reid WD. Influence of inspiratory muscle weakness on inspiratory muscle training responses in chronic heart failure patients: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2014 Jul;95(7):1398-407. doi: 10.1016/j.apmr.2014.02.022. Epub 2014 Mar 13. PMID 24631801
- [Background] Russo N, Compostella L, Tarantini G, Setzu T, Napodano M, Bottio T, D'Onofrio A, Isabella G, Gerosa G, Iliceto S, Bellotto F. Cardiac rehabilitation after transcatheter versus surgical prosthetic valve implantation for aortic stenosis in the elderly. Eur J Prev Cardiol. 2014 Nov;21(11):1341-8. doi: 10.1177/2047487313494029. Epub 2013 Jun 11. PMID 23757283
- [Background] Voller H, Salzwedel A, Nitardy A, Buhlert H, Treszl A, Wegscheider K. Effect of cardiac rehabilitation on functional and emotional status in patients after transcatheter aortic-valve implantation. Eur J Prev Cardiol. 2015 May;22(5):568-74. doi: 10.1177/2047487314526072. Epub 2014 Feb 27. PMID 24577878
- [Background] Fauchere I, Weber D, Maier W, Altwegg L, Luscher TF, Grunenfelder J, Nowak A, Tuller D, Genoni M, Falk V, Hermann M. Rehabilitation after TAVI compared to surgical aortic valve replacement. Int J Cardiol. 2014 May 15;173(3):564-6. doi: 10.1016/j.ijcard.2014.03.121. Epub 2014 Mar 21. No abstract available. PMID 24713461
- [Background] Sbruzzi G, Ribeiro RA, Schaan BD, Signori LU, Silva AM, Irigoyen MC, Plentz RD. Functional electrical stimulation in the treatment of patients with chronic heart failure: a meta-analysis of randomized controlled trials. Eur J Cardiovasc Prev Rehabil. 2010 Jun;17(3):254-60. doi: 10.1097/HJR.0b013e328339b5a2. PMID 20560163